CLINICAL TRIAL: NCT00343018
Title: Evaluating the NICHD Interview Protocol in an Analog Study
Brief Title: Interviewing Children About Past Events: Evaluating the NICHD Interview Protocol
Status: Completed | Type: Observational
Sponsor: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999904108; 04-CH-N108
Record Dates: First submitted 2006-06-19; First posted 2006-06-21 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2006-10-05

CONDITIONS: Memory
Keywords: Preschoolers; Young Children; Eyewitness; Memory

SUMMARY:
This study, conducted by the NICHD in collaboration with Lancaster University in Lancaster, England, will evaluate the accuracy of information obtained from children using AN ADAPTED VERSION OF NICHD's interview protocol. The NICHD protocol was developed to help forensic interviewers OBTAIN INFORMATION FROM children who may be victims of or witnesses to a crime ABOUT THEIR EXPERIENCES. This study does not involve forensic interviews, but is DESIGNED TO OBTAIN INFORMATION FROM children ABOUT an event that takes place at their school. The study will examine how children report a brief interaction with an unfamiliar adult, how the memory of the event changes over time, and how the use of different interview techniques can help children give a fuller and more accurate accounts of past experiences.

Children 5 and 6 years of age who attend local schools in the Lancaster, England, area may be eligible for this study. Participants will be told that they are going to have their pictures taken and will be escorted by a researcher to a room at the school with another researcher who is posing as a photographer. The "photographer" and the child will put on a costume, such as a pirate's outfit, over their street clothes, helping each other put on pieces of the costume. The photographer will take pictures of the child in the costume. They will each take off the costumes and the child will be told that he or she will receive the photographs at a later time. Another researcher posing as a photographer will come into the room, interrupting the event, and begin to argue with the first photographer about who had booked the equipment. They will resolve the argument and apologize to the child for the interruption.

About 6 weeks after the event, the children will be interviewed using the ADAPTED VERSION OF NICHD interview protocol. Half will be interviewed first about the staged event (the photo session), followed by an interview about a fictitious event (e.g., a class visit to the fire station) that could plausibly have happened but did not. The other half of the children will be interviewed first about the fictitious event and then about the staged event. The children will be interviewed according to one of the following three procedures:

* The NICHD protocol preceded by a rapport-building phase that includes the rules of the interview and open-ended questions about the child and a recently experienced event
* The NICHD protocol preceded by a rapport-building phase that includes the rules of the interview and direct questions about the child and a recently experienced event, or
* The NICHD protocol preceded by the rules of the interview and open-ended questions about the child, but no opportunity to practice talking about a recently experienced event.

After the interviewer has elicited as much information as is likely to be gained from verbal questions, he or she will present the child with a line drawing of a gender neutral person and ask the child to indicate where the child was touched by the photographer and where the child touched the photographer. Any child who provides a report of the fictitious event will be interviewed in the same way about the fictitious event. After 1 year, the children will be interviewed again in the same manner as the 6-week interview.

The interviews will be audio- and videotaped to record the kind of information the children talk about and compare it to what actually happened in the event.

DETAILED DESCRIPTION:
The NICHD interview protocol was designed to aid forensic interviewers in adhering to best standards of practice when interviewing children. Field studies evaluating its use have demonstrated improvements in both interviewer behavior, and the amount and quality of information obtained from children, compared to interviews conducted prior to its implementation in test sites. Because field studies were conducted in forensic settings, however, it has not been possible to evaluate the protocol's effect on the accuracy of information reported by children. This present study therefore aims to evaluate the accuracy of information obtained using the NICHD interview protocol in an analog study. In addition the study is designed to explore children's willingness to provide details of a suggested, non-experienced event, and the effectiveness of including a human figure drawing as an auxiliary technique for eliciting further information. Furthermore, we will explore the importance of the pre-substantive/rapport-building phase of interviews, and the impact this has on children's reports of experienced and suggested events. Finally, we will explore the effectiveness of the interview protocol with children when a long delay has occurred between the event and the interview.

Children will take part, individually, in a staged event at their school, and approximately six weeks later, be interviewed at the university about what they experienced. In addition, children will be asked to talk about a suggested fictitious event (one that has not happened). The order of the interviews will be counter-balanced across children and rapport-building conditions. Some children will be interviewed with an open-ended script that includes practice in episodic memory, some with a script made up of direct questions, including a practice in episodic memory, and some with one that uses open-ended questions but does not provide practice in talking about an event from episodic memory. Approximately one year later children will be interviewed again, so that we can examine children's reports in protocol interviews over a long delay. Children's reports will be analyzed for both overall amount and accuracy of information reported, as well as in response to the different cues and props given in the course of the interview. It is not anticipated that the study will pose any risks to the children involved, and we expect that both the staged event and the interviews will be enjoyable and stimulating. We expect that the results of the study will provide further support for the use of NICHD interview as a safe and effective means of interviewing children about past experiences. In addition to general information on children's eyewitness capabilities, the study is expected to supplement field studies by contributing knowledge about the accuracy of children's memory using the NICHD interview protocol.

ELIGIBILITY:
* INCLUSION CRITERIA:

Children between the ages of 5-6.

All children within the nominated age range attending the participating schools, whose parents have given consent, will be included in the study.

If children are identified as having specific disabilities that may affect their abiity to give a report about their experience (e.g., a developmental delay), or if English is a second language and inadequate mastery at the time of interview affects the child's reports, they will be included in the event and interviewed, but their data will be excluded from later analysis.

Min Age: 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 150
Dates: Start 2004-01-21; Study Completion 2006-10-05

CONTACTS AND LOCATIONS:
Locations (1):
- National Institute of Child Health and Human Development (NICHD), Bethesda, Maryland, United States

REFERENCES:
- [Background] Ceci SJ, Bruck M. Suggestibility of the child witness: a historical review and synthesis. Psychol Bull. 1993 May;113(3):403-39. doi: 10.1037/0033-2909.113.3.403. PMID 8316609